CLINICAL TRIAL: NCT01089062
Title: A Randomized, Double Blind, Placebo Controlled, Three-Period Crossover Study Comparing the Acute Effects of Intravenous Dihydroergotamine (DHE) and Orally Inhaled DHE (MAP0004) on Pulmonary Arterial Pressure and Tolerability in Healthy Adults
Brief Title: Pharmacodynamic Study to Compare Acute Effects of Dihydroergotamine Mesylate (DHE) on Pulmonary Arterial Pressure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Collaborators: MAP Pharmaceuticals, Inc., a wholly owned subsidiary of Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MAP0004-CL-P102
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Results first posted 2013-10-22 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: Healthy volunteers
MeSH Terms: interventions — Sodium Chloride; Dihydroergotamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment A, then Treatment B, then Treatment C (Other): The second dose in each treatment group (A,B,C) was given two hours from the time of the first dose. There were 7-11 days between each treatment visit.
  Treatment A = inhaler placebo and IV DHE for first dose, inhaler placebo for second dose at Visit 2.
  Treatment B = MAP0004 1.0mg and IV placebo for first dose, MAP0004 1.0mg for second dose at Visit 3.
  Treatment C = inhaler placebo and IV placebo for first dose, inhaler placebo for second dose at Visit 4.
  Interventions: Drug: MAP0004; Drug: IV Placebo (Saline); Drug: Placebo Inhaler; Drug: IV Dihydroergotamine Mesylate (DHE)
- Treatment A, then Treatment C, then Treatment B (Other): The second dose in each treatment group (A,C,B) was given two hours from the time of the first dose. There were 7-11 days between each treatment visit.
  Treatment A = inhaler placebo and IV DHE for first dose, inhaler placebo for second dose at Visit 2.
  Treatment C = inhaler placebo and IV placebo for first dose, inhaler placebo for second dose at Visit 3.
  Treatment B = MAP0004 1.0mg and IV placebo for first dose, MAP0004 1.0mg for second dose at Visit 4.
  Interventions: Drug: MAP0004; Drug: IV Placebo (Saline); Drug: Placebo Inhaler; Drug: IV Dihydroergotamine Mesylate (DHE)
- Treatment B, then Treatment A, then Treatment C (Other): The second dose in each treatment group (B,A,C) was given two hours from the time of the first dose. There were 7-11 days between each treatment visit.
  Treatment B = MAP0004 1.0mg and IV placebo for first dose, MAP0004 1.0mg for second dose at Visit 2.
  Treatment A = inhaler placebo and IV DHE for first dose, inhaler placebo for second dose at Visit 3.
  Treatment C = inhaler placebo and IV placebo for first dose, inhaler placebo for second dose at Visit 4.
  Interventions: Drug: MAP0004; Drug: IV Placebo (Saline); Drug: Placebo Inhaler; Drug: IV Dihydroergotamine Mesylate (DHE)
- Treatment B, then Treatment C, then Treatment A (Other): The second dose in each treatment group (B,C,A) was given two hours from the time of the first dose. There were 7-11 days between each treatment visit.
  Treatment B = MAP0004 1.0mg and IV placebo for first dose, MAP0004 1.0mg for second dose at Visit 2.
  Treatment C = inhaler placebo and IV placebo for first dose, inhaler placebo for second dose at Visit 3.
  Treatment A = inhaler placebo and IV DHE for first dose, inhaler placebo for second dose at Visit 4.
  Interventions: Drug: MAP0004; Drug: IV Placebo (Saline); Drug: Placebo Inhaler; Drug: IV Dihydroergotamine Mesylate (DHE)
- Treatment C, then Treatment A, then Treatment B (Other): The second dose in each treatment group (C,A,B) was given two hours from the time of the first dose. There were 7-11 days between each treatment visit.
  Treatment C = inhaler placebo and IV placebo for first dose, inhaler placebo for second dose at Visit 2.
  Treatment A = inhaler placebo and IV DHE for first dose, inhaler placebo for second dose at Visit 3.
  Treatment B = MAP0004 1.0mg and IV placebo for first dose, MAP0004 1.0mg for second dose at Visit 4.
  Interventions: Drug: MAP0004; Drug: IV Placebo (Saline); Drug: Placebo Inhaler; Drug: IV Dihydroergotamine Mesylate (DHE)
- Treatment C, then Treatment B, then Treatment A (Other): The second dose in each treatment group (C,B,A) was given two hours from the time of the first dose. There were 7-11 days between each treatment visit.
  Treatment C = inhaler placebo and IV placebo for first dose, inhaler placebo for second dose at Visit 2.
  Treatment B = MAP0004 1.0mg and IV placebo for first dose, MAP0004 1.0mg for second dose at Visit 3.
  Treatment A = inhaler placebo and IV DHE for first dose, inhaler placebo for second dose at Visit 4.
  Interventions: Drug: MAP0004; Drug: IV Placebo (Saline); Drug: Placebo Inhaler; Drug: IV Dihydroergotamine Mesylate (DHE)

INTERVENTIONS:
Drug: MAP0004 — 1.0 mg orally inhaled MAP0004 administered in Treatment B as per protocol
Drug: IV Placebo (Saline) — IV Placebo (Saline) administered in Treatment B and Treatment C as per protocol
Drug: Placebo Inhaler — Orally inhaled Placebo administered in Treatment A and Treatment C as per protocol.
Drug: IV Dihydroergotamine Mesylate (DHE) — IV DHE administered in Treatment A as per protocol
  Other Names: D.H.E.45®

SUMMARY:
Compare the acute effects and tolerability of Dihydroergotamine Mesylate (DHE) delivered by Oral Inhalation (MAP0004) versus by intravenous (IV) infusion in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide a signed, executed written informed consent
2. Healthy non-smoking adult volunteers: Male or Female subjects 18 to 45 years old
3. Female subjects who are practicing adequate contraception
4. Stable cardiac status
5. Normal hemoglobin values
6. Normal Echocardiogram
7. Normal or not clinically significant 12-lead Electrocardiogram
8. Demonstrated ability to properly use the Tempo® Inhaler
9. Subject has not donated blood in the last 56 days

Exclusion Criteria:

1. Contraindication to dihydroergotamine mesylate (DHE)
2. Use of any excluded concomitant medications within the 10 days prior to Visit 1
3. History of hemiplegic or basilar migraine
4. Participation in another investigational trial during the 30 days prior to Visit 1

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Noveck, M.D., Ph.D., Principal Investigator — Duke Clinical Research Unit
Locations (1):
- Duke Clinical Research Unit, Durham, North Carolina, United States

REFERENCES:
- [Derived] Noveck RJ, Douglas PS, Chow SC, Mangum B, Kori S, Kellerman DJ. Assessing acute systemic effects of an inhaled drug with serial echocardiography: a placebo-controlled comparison of inhaled and intravenous dihydroergotamine. Drug Des Devel Ther. 2013 Jul 24;7:619-25. doi: 10.2147/DDDT.S44093. Print 2013. PMID 23926420

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a 3-treatment, 3-period, 6-sequence crossover study. Each subject received all 3 treatments in a randomly assigned order: treatments A, B, and C, the sequences were ABC, ACB, BAC, BCA, CAB, and CBA.
Groups:
- Treatment A, Then B, Then C: The second dose in each treatment group (A,B,C) was given two hours from the time of the first dose. There were 7-11 days between each treatment visit.
  Treatment A = inhaler placebo and Intravenous (IV) Dihydroergotamine (DHE) for first dose, inhaler placebo for second dose at Visit 2.
  Treatment B = MAP0004 1.0mg and IV placebo for first dose, MAP0004 1.0mg for second dose at Visit 3.
  Treatment C = inhaler placebo and IV placebo for first dose, inhaler placebo for second dose at Visit 4.
- Treatment A, Then C, Then B: The second dose in each treatment group (A,C,B) was given two hours from the time of the first dose. There were 7-11 days between each treatment visit.
  Treatment A = inhaler placebo and IV DHE for first dose, inhaler placebo for second dose at Visit 2.
  Treatment C = inhaler placebo and IV placebo for first dose, inhaler placebo for second dose at Visit 3.
  Treatment B = MAP0004 1.0mg and IV placebo for first dose, MAP0004 1.0mg for second dose at Visit 4.
- Treatment B, Then A, Then C: The second dose in each treatment group (B,A,C) was given two hours from the time of the first dose. There were 7-11 days between each treatment visit.
  Treatment B = MAP0004 1.0mg and IV placebo for first dose, MAP0004 1.0mg for second dose at Visit 2.
  Treatment A = inhaler placebo and IV DHE for first dose, inhaler placebo for second dose at Visit 3.
  Treatment C = inhaler placebo and IV placebo for first dose, inhaler placebo for second dose at Visit 4.
- Treatment B, Then C, Then A: The second dose in each treatment group (B,C,A) was given two hours from the time of the first dose. There were 7-11 days between each treatment visit.
  Treatment B = MAP0004 1.0mg and IV placebo for first dose, MAP0004 1.0mg for second dose at Visit 2.
  Treatment C = inhaler placebo and IV placebo for first dose, inhaler placebo for second dose at Visit 3.
  Treatment A = inhaler placebo and IV DHE for first dose, inhaler placebo for second dose at Visit 4.
- Treatment C, Then A, Then B: The second dose in each treatment group (C,A,B) was given two hours from the time of the first dose. There were 7-11 days between each treatment visit.
  Treatment C = inhaler placebo and IV placebo for first dose, inhaler placebo for second dose at Visit 2.
  Treatment A = inhaler placebo and IV DHE for first dose, inhaler placebo for second dose at Visit 3.
  Treatment B = MAP0004 1.0mg and IV placebo for first dose, MAP0004 1.0mg for second dose at Visit 4.
- Treatment C, Then B, Then A: The second dose in each treatment group (C,B,A) was given two hours from the time of the first dose. There were 7-11 days between each treatment visit.
  Treatment C = inhaler placebo and IV placebo for first dose, inhaler placebo for second dose at Visit 2.
  Treatment B = MAP0004 1.0mg and IV placebo for first dose, MAP0004 1.0mg for second dose at Visit 3.
  Treatment A = inhaler placebo and IV DHE for first dose, inhaler placebo for second dose at Visit 4.
Period: Visit 2 (Randomization)
Arm/Group | Treatment A, Then B, Then C | Treatment A, Then C, Then B | Treatment B, Then A, Then C | Treatment B, Then C, Then A | Treatment C, Then A, Then B | Treatment C, Then B, Then A
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 3 | 3 | 3 | 4 | 3 | 3
Not Completed | 1 | 1 | 1 | 0 | 1 | 1
Period: Visit 3
Arm/Group | Treatment A, Then B, Then C | Treatment A, Then C, Then B | Treatment B, Then A, Then C | Treatment B, Then C, Then A | Treatment C, Then A, Then B | Treatment C, Then B, Then A
Started | 3 | 3 | 3 | 4 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Period: Visit 4
Arm/Group | Treatment A, Then B, Then C | Treatment A, Then C, Then B | Treatment B, Then A, Then C | Treatment B, Then C, Then A | Treatment C, Then A, Then B | Treatment C, Then B, Then A
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Follow-up Visit (Final Visit)
Arm/Group | Treatment A, Then B, Then C | Treatment A, Then C, Then B | Treatment B, Then A, Then C | Treatment B, Then C, Then A | Treatment C, Then A, Then B | Treatment C, Then B, Then A
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment A, Then B, Then C; Treatment A, Then C, Then B; Treatment B, Then A, Then C; Treatment B, Then C, Then A; Treatment C, Then A, Then B; Treatment C, Then B, Then A: Treatment A = inhaler placebo and IV DHE for first dose, inhaler placebo for second dose.
  Treatment B = MAP0004 1.0mg and IV placebo for first dose, MAP0004 1.0mg for second dose.
  Treatment C = inhaler placebo and IV placebo for first dose, inhaler placebo for second dose.
- Total: Total of all reporting groups
Arm/Group | Treatment A, Then B, Then C | Treatment A, Then C, Then B | Treatment B, Then A, Then C | Treatment B, Then C, Then A | Treatment C, Then A, Then B | Treatment C, Then B, Then A | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.6 (9.2) | 23.4 (3.9) | 28.2 (8.2) | 30.3 (4.7) | 26.5 (7.4) | 24.8 (7.2) | 26.6 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 2 | 4 | 1 | 3 | 16
  Male | 2 | 0 | 2 | 0 | 3 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-2hrs) of Pulmonary Arterial Systolic Pressure (PASP) Over Time Post 1st Dose
Description: AUC(0-2hrs) (Area Under the Curve, time 0-2 hours post-1st dose) in PASP millimeters of mercury times minutes (mmHg*min). PASP is the highest pressure exerted on the walls of the pulmonary artery.
Time Frame: 2 hours from time of first dose
Population: Patients with available data at the required time point were included in the analysis population.
Measure: Mean (Standard Deviation); unit: mmHg*min
Groups:
- Treatment A: Treatment A = inhaler placebo and IV DHE for first dose, inhaler placebo for second dose.
- Treatment B: Treatment B = MAP0004 1.0mg and IV placebo for first dose, MAP0004 1.0mg for second dose.
- Treatment C: Treatment C = inhaler placebo and IV placebo for first dose, inhaler placebo for second dose.
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 18 | 18 | 18
mmHg*min | 2794.93 (476.66) | 2580.06 (389.06) | 2497.71 (384.29)

2. Secondary Outcome: Percent of Subjects With an Increase in PASP Greater Than 10mmHg From Baseline to 2 Hours From the First Dose
Description: Pulmonary artery systolic pressure (PASP) is the highest pressure exerted on the walls of the pulmonary artery.
Time Frame: baseline and 2 hours from the time of first dose
Population: Patients with available data at the required time point were included in the analysis population.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 24 | 24 | 24
percentage of participants | 4.2 | 0.0 | 0.0

3. Secondary Outcome: Maximum Change in PASP From Baseline to the Two Hour Period Following the First Dose
Description: Pulmonary artery systolic pressure (PASP) is the highest pressure exerted on the walls of the pulmonary artery.
Time Frame: baseline and 2 hours from the time of first dose
Population: Patients with available data at the required time point were included in the analysis population.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 24 | 24 | 24
mmHg
  Baseline | 22.8 (4.4) | 19.2 (4.6) | 21.2 (3.3)
  Max Change from Baseline over 2 hrs from 1st dose | 7.8 (2.4) | 6.1 (2.8) | 4.0 (1.7)

4. Secondary Outcome: AUC(0-4hrs) of Pulmonary Arterial Systolic Pressure (PASP) From the Start of the First Dose to Two Hours After the Second Dose
Description: AUC(0-4hrs) (Area Under the Curve, time 0-4 hours post-1st dose) in PASP millimeters of mercury times minutes (mmHg*min). PASP is the highest pressure exerted on the walls of the pulmonary artery.
Time Frame: 4 hours from the time of first dose
Population: Patients with available data at the required time point were included in the analysis population.
Measure: Mean (Standard Deviation); unit: mmHg*min
Groups:
- Treatment A: Treatment A = inhaler placebo and IV DHE for first dose, inhaler placebo for second dose 2 hours from time of first dose.
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 24 | 24 | 24
mmHg*min | 5700.11 (1016.86) | 5336.38 (823.51) | 4907.03 (773.11)

5. Secondary Outcome: Change in Blood Pressure From Baseline After the Two 2-hour Post Dosing Periods
Description: Systolic and diastolic blood pressure measure the lowest and highest pressures against the walls of the arteries. Changes were calculated from 30 minutes pre dose (baseline) to 10 minutes post first and second dose. A positive change from baseline indicates an increase in blood pressure and a negative change indicates a decrease in blood pressure.
Time Frame: baseline, 10 minutes post 1st dose, 10 minutes post 2nd dose
Population: Patients with available data at the required time point were included in the analysis population.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 20 | 20 | 20
mmHg
  Baseline Systolic | 112.5 (11.3) | 113.3 (15.3) | 113.2 (12.3)
  Change at 10 min in Systolic after 1st dose | 10.4 (10.0) | 4.7 (8.5) | 0.4 (7.9)
  Change at 10 min in Systolic after 2nd dose | 0.2 (7.8) | 1.2 (9.9) | -0.5 (5.2)
  Baseline Diastolic | 65.8 (7.3) | 67.2 (9.1) | 64.4 (6.7)
  Change at 10 min in Diastolic after 1st dose | 7.0 (7.2) | 2.0 (8.0) | 1.1 (5.1)
  Change at 10 min in Diastolic after 2nd dose | -1.5 (11.2) | -2.0 (9.4) | 0.1 (4.9)

6. Secondary Outcome: Change From Baseline in QTc Interval at 14 Minutes After the 1st and 2nd Dose
Description: The corrected QT interval (QTc) is a measurement of the electrical impulses through the largest part of the heart muscle. A negative change is a shortening of the QTc interval, a positive change is a lengthening of the QTc interval.
Time Frame: baseline, 14 minutes from time of 1st dose, 14 minutes from time of 2nd dose
Population: Patients with available data at the required time point were included in the analysis population.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 20 | 20 | 20
milliseconds
  Baseline | 403.9 (15.8) | 402.3 (19.0) | 399.9 (16.4)
  Change from baseline at 14 mins post 1st dose | -5.8 (12.2) | -0.8 (5.6) | 2.4 (10.8)
  Change from baseline at 14 mins post 2nd dose | 1.5 (10.7) | -0.8 (13.4) | 4.1 (9.6)

ADVERSE EVENTS:
Description: All subjects who were randomized and received at least one dose of study drug were included in the adverse event analysis. Adverse events are presented by treatment arm, not by individual treatment (intervention) received.
Arm/Group | Treatment A | Treatment B | Treatment C
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 19/20 | 10/20 | 6/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=20) | Treatment B (N=20) | Treatment C (N=20)
Headache (Nervous system disorders) | 6 | 5 | 1
Dizziness (Nervous system disorders) | 3 | 2 | 1
Burning sensation (Nervous system disorders) | 4 | 0 | 0
Paraesthesia (Nervous system disorders) | 3 | 0 | 0
Head discomfort (Nervous system disorders) | 2 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 0
Sensory Disturbance (Nervous system disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 10 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Feeling hot (General disorders) | 8 | 0 | 0
Chest discomfort (General disorders) | 2 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Infusion site pain (General disorders) | 0 | 1 | 0
Sensation of pressure (General disorders) | 1 | 0 | 0
Pharmaceutical product complaint (Social circumstances) | 4 | 2 | 1 — Medication Aftertaste
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 2 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Heart rate increased (Investigations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.